CLINICAL TRIAL: NCT04366492
Title: Prevalence of Blood Borne Viral Infections (HBV/HCV/HIV) in the Belgian Prison System
Brief Title: HBV/HCV/HIV in Belgian Prisons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HBV-HCV-HIV-001
Record Dates: First submitted 2020-02-05; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis C; Hepatitis B; HIV Infections
MeSH Terms: conditions — Hepatitis C; Hepatitis B; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- persons in prison (Other)
  Interventions: Other: Prevalence of blood borne viral infections (HBV/HCV/HIV)

INTERVENTIONS:
Other: Prevalence of blood borne viral infections (HBV/HCV/HIV) — rapid finger prick test for HCV Ab, HBsAg and HIV and a questionnaire

SUMMARY:
To assess the prevalence of blood-borne viral infections in prisons in Belgium, screening will be executed in several prisons in Flanders, Brussels and Wallonia to obtain a geographical representative distribution.

Upon informed consent screening will be performed using whole capillary blood (finger prick testing) with three different tests for HCV Ab, HBsAg and HIV. Screening will be performed first. While awaiting the test result (15-20min), the participant can fill out a questionnaire (together with the study nurse), concerning risk factors for HCV, HBV and HIV infection. This questionnaire is filled out directly online, and will be immediately implemented in the encoded database. The database is set-up according to the rules of good clinical practice. (Castor EDC software). The results will be filled out immediately by the prison staff in this database after it is filled out by the participant, minimizing the risk of displacement of test results.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Imprisoned in one of the predefined prisons in Flanders Brussels or Wallonia participating in this trial
* Written informed consent obtained

Exclusion Criteria:

* Written informed consent not possible: (language barrier, illiteracy)
* Already participated in the study: re-entry within inclusion period in one of the prisons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3045 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with HCV Ab+ (Hepatitis C Virus Antibody) | day 1
  test using whole capillary blood (finger prick testing)
Number of participants with HBsAg+ (Hepatitis B surface Antigen) | day 1
  test using whole capillary blood (finger prick testing)
Number of participants with HIV Ab+ (human immunodeficiency virus antibody) | day1
  test using whole capillary blood (finger prick testing)

SECONDARY OUTCOMES:
.Prevalence of blood-borne viral infections in Belgian prisons | day 1
  number of HCV Ab+/number of screened prisoners by finger prick
  * number of HBsAg+/number of screened prisoners by finger prick
  * number of HIV Ab+/number of screened prisoners by finger prick
5. Questionnaire to Identify risk factors associated with the aforementioned blood borne viral infections (hepatitis C, hepatitis B and HIV) in prison | day 1
  i. Combine results from positive finger prick test with questionnaire regarding sociodemographic factors, migration, risk factors for blood born viruses (sexual contacts, incarceration, drug use)
Analysis of uptake counselling by physician in prison | day 1
  Percentage of patients with a positive finger prick test who attend a consultation by the prison physician in relation of total tested positive on finger prick
Analysis of uptake of anti(retro)viral treatment | day 1
  percentage of positive clients who started treatment in relation of total of positive clients needing treatment

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, MD, PhD, Principal Investigator — Hasselt University; Dana Busschots, drs., Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - UZ Gent, Ghent
  - Hasselt University, Hasselt

REFERENCES:
- [Derived] Busschots D, Kremer C, Bielen R, Koc OM, Heyens L, Brixko C, Laukens P, Orlent H, Bilaey P, De Smet F, Hellemans G, Muyldermans G, Van Baelen L, Hens N, Van Vlierberghe H, Robaeys G. A multicentre interventional study to assess blood-borne viral infections in Belgian prisons. BMC Infect Dis. 2021 Jul 27;21(1):708. doi: 10.1186/s12879-021-06405-z. PMID 34315415